CLINICAL TRIAL: NCT03275818
Title: Phase II Trial of Nab-paclitaxel for the Treatment of Desmoid Tumors and Multiply Relapsed/Refractory Desmoplastic Small Round Cell Tumors and Ewing Sarcoma
Brief Title: Trial of Nab-paclitaxel in Patients With Desmoid Tumors and Multiply Relapsed/Refractory Desmoplastic Small Round Cell Tumors and Ewing Sarcoma
Acronym: ABRADES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-39; 2016-002464-14 (EudraCT Number)
Record Dates: First submitted 2017-08-03; First posted 2017-09-08 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-04

CONDITIONS: Tumor, Desmoplastic Small Round Cell, Adult; Tumor, Desmoplastic Small Round Cell, Childhood; Sarcoma, Ewing; Sarcoma; Desmoid
Keywords: sarcoma; Desmoid tumor; Desmoplastic small round cell tumor; Ewing sarcoma; relapsed; refractory
MeSH Terms: conditions — Neoplasms; Sarcoma, Ewing; Sarcoma; Desmoid Tumors; Desmoplastic Small Round Cell Tumor; Recurrence | interventions — Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel (Experimental): nab-paclitaxel (ABRAXANE) will be administered as follows:
  * Age ≥ 21: 125 mg/m2 days 1, 8 and 15 in cycles of 28 days
  * Age ≥ 6 months and ≤ 20 years: 240 mg/m2 (for patients weighing > 10 kg) and 11.5 mg/kg (for patients weighing ≤ 10 kg) on days 1, 8 and 15 in cycles of 28 days
  Interventions: Drug: nab paclitaxel

INTERVENTIONS:
Drug: nab paclitaxel — Subjects in the DT cohort will receive a maximum of three cycles. Subjects in the DSRCT and ES cohort will receive unlimited cycles until disease progression, the subject begins a new anticancer treatment, withdrawal of parent/guardian/subject consent/assent, parent/guardian/subject refusal, physician decision, toxicity that cannot be managed by dose delay or dose reduction alone or the study ends for any reason
  Other Names: Abraxane

SUMMARY:
A two-cohort, fase II, open-label, non-randomized, multicenter clinical trial. 14 sites in Spain.

Cohort 1: Subjects with desmoid tumor (DT) Cohort 2: Subjects with desmoplastic small round cell tumor or Ewing sarcoma (DSRCT and ES)

Nab-paclitaxel (ABRAXANE) will be administered as follows:

Age ≥ 21 and ≤ 80 years: 125 mg/m2 days 1, 8 and 15 in cycles of 28 days Age ≥ 6 months and ≤ 20 years: 240 mg/m2 days 1, 8 and 15 in cycles of 28 days

Subjects in the DT cohort will receive a maximum of three cycles. Subjects in the DSRCT and ES cohort will receive unlimited cycles until disease progression, the subject begins a new anticancer treatment, withdrawal of parent/guardian/subject consent/assent, parent/guardian/subject refusal, physician decision, toxicity that cannot be managed by dose delay or dose reduction alone or the study ends for any reason.

The main goal is to determine the objective response rate (ORR), using RECIST 1.1 criteria and to determine the clinical benefit rate (CBR), defined as CR+PR+SD for 3 months with improvement of pain with at least minimally important difference (MID) of 2 in subjects with desmoid tumors (DT cohort) and to determine the objective response rate (ORR) in subjects with desmoplastic small round cell tumor and Ewing sarcoma, using RECIST 1.1 criteria (DSRCT and ES cohort)

ELIGIBILITY:
TD Cohort

Inclusion Criteria:

1. Subjects (parent or legal guardian if subject under 18 years) must voluntarily sign the informed consent form before any study test is conducted that is not part of routine subject care.
2. Subjects with pathologic diagnosis of deep desmoid tumor of extremities, trunk wall or head and neck region.Intra-abdominal desmoid tumor cases could be enrolled if harboring betacatenin mutation.
3. Subjects must be symptomatic (pain) due to tumor desmoid mass or lack physical function due to desmoid tumor mass, or in RECIST progression in the last 6 months.
4. Age: ≥ 6 months.
5. Subjects could have received one previous chemotherapy line if the scheme was methotrexate plus vinca alkaloids. Patients who received prostaglandin inhibitors or hormone therapy are also eligible.
6. Availability of archive tumor block.
7. Measurable disease, according to RECIST 1.1 criteria.
8. Performance status ≤1 (ECOG).
9. Normal ECG values.
10. Adequate bone marrow function (hemoglobin ≥ 9 g/dL, leukocytes ≥ 3.000/mm3, neutrophils ≥ 1.500/mm3, platelets ≥ 100.000/mm3). Subjects with plasma creatinine ≤ 1.6 mg/dl, transaminases ≤ 2.5 times the ULN, total bilirubin ≤ 1.25 times the ULN are acceptable.
11. Men or women of childbearing potential must use an effective method of contraception before entry into the study and throughout the same and for 6 months after ending the study treatment. Women of childbearing potential must have a negative urine or serum pregnancy test before study entry.
12. HBV and HCV serologies must be performed prior to inclusion. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA VHB+) remaining at investigators' discretion the preventive treatment with lamivudine. If a potential subject is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the subject should NOT be included in the study (if a qualitative PCR cannot be performed then subject will not be able to enter the study).

Exclusion Criteria:

1. Prior taxane therapy for any indication.
2. Less than 4 weeks elapsed since prior exposure to chemotherapy.
3. More than one previous chemotherapy line.
4. Subjects with desmoid tumor of abdominal cavity (abdominal wall is not an exclusion criterion)
5. Desmoid tumor with ill-defined margins.
6. Unavailability to undergo MRI.
7. Previously irradiated target lesion (if radiation dose exceeded 50 Gy).
8. Pre-existing neuropathy greater than grade 1.
9. Other active invasive malignancy requiring ongoing therapy or expected to require systemic therapy within two years. However, localized squamous cell carcinoma of the skin, basal cell carcinoma of the skin, carcinoma in situ of the cervix or other malignancies requiring only locally ablative therapy, will not result in exclusion.
10. Concomitant anticancer therapy, immunotherapy or radiation therapy within prior 4 weeks.
11. Uncontrolled intercurrent illness including but not limited to ongoing or active infection requiring IV antibiotic, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness or social situations that would limit compliance with study requirements
12. Hb < 9 g/dL.
13. Women who are pregnant or breast-feeding.
14. Known hypersensitivity to protein bound paclitaxel
15. Any other concurrent condition that in the investigators opinion would jeopardize compliance with the protocol
16. Known positive test for infection by human immunodeficiency virus (HIV).
17. Subjects participating in another clinical trial or receiving any other investigational product.

DSRCT and ES Cohort

Inclusion Criteria:

1. Subjects or legal guardian must voluntarily sign the informed consent form before any study test is conducted that is not part of routine subject care.
2. Subject diagnosed of relapsed/refractory desmoplastic small round cell tumor (DSRCT) or Ewing´s sarcoma.
3. DSRCT subjects must have received at least one previous poli-chemotherapy line.
4. Ewing´s sarcoma subjects must have received at least two standard chemotherapy lines.
5. Age ≥ 6 months
6. Availability of archive tumor blocks or slides (new biopsy recommended).
7. Measurable disease, according to RECIST 1.1 criteria.
8. Performance status ≤1 (ECOG).
9. Adequate respiratory functions: FEV1 > 1L.
10. Normal ECG values.
11. Adequate bone marrow function (hemoglobin ≥ 9 g/dL, leukocytes ≥ 3,000/mm3, neutrophils ≥ 1,500/mm3, platelets ≥ 100,000/mm3). Subjects with plasma creatinine ≤ 1.6 mg/dL, transaminases ≤ 2.5 times the ULN, total bilirubin ≥ 1.25 times ULN, CPK ≤ 2.5 times ULN, alkaline phosphatase ≤ 2.5 times the ULN are acceptable. If alkaline phosphatase is > 2.5 times the ULN, then the alkaline phosphatase liver fraction and/or 5' nucleotidase and/or GGT must be ≤ ULN.
12. Men or women of child bearing potential should be using an effective method of contraception before entry into the study and throughout the same and for 6 months after ending the study. Women of childbearing potential must have a negative urine pregnancy test before study entry.
13. HBV and HCV serologies must be performed prior to inclusion. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA VHB+) remaining at investigators' discretion the preventive treatment with lamivudine. If a potential subject is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the subject should NOT be included in the study (if a qualitative PCR cannot be performed then subject will not be able to enter the study).
14. Prior taxane therapy for any indication is accepted.
15. > Grade 3 (intense and diffuse) expression of SPARC by immunohistochemistry.

Exclusion criteria:

1. Less than 4 weeks elapsed since prior exposure to chemotherapy.
2. Pre-existing neuropathy greater than Grade 1.
3. Other active invasive malignancy requiring ongoing therapy or expected to require systemic therapy within two years. However, localized squamous cell carcinoma of the skin, basal cell carcinoma of the skin, carcinoma in situ of the cervix or other malignancies requiring only locally ablative therapy, will not result in exclusion.
4. Concomitant anticancer therapy, immunotherapy or radiation therapy within prior 4 weeks.
5. Uncontrolled intercurrent illness including but not limited to ongoing or active infection requiring IV antibiotic, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness or social situations that would limit compliance with study requirements
6. Hb < 9 g/dL.
7. Women who are pregnant or breast-feeding.
8. Known hypersensitivity to protein bound paclitaxel.
9. Any other concurrent condition that in the investigators opinion would jeopardize compliance with the protocol.
10. Known positive test for infection by human immunodeficiency virus (HIV).
11. Subjects participating in another clinical trial or receiving any other investigational product.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) - cohort 1 | 3 months
  TD cohort: Overall response rate (ORR) according to RECIST 1.1 and/or clinical benefit rate (CBR) at 3 months with pain improvement of at least 2 points in the Brief Pain Inventory - Short Form (BPI-SF)
Objective response rate (ORR) - cohort 2 | 2 months
  DSRCT and SE cohort: To determine the objective response rate (ORR) in subjects with desmoplastic small round cell tumor and Ewing's sarcoma, using RECIST 1.1 criteria

SECONDARY OUTCOMES:
Pattern of radiological response - cohort 1 | 3 months
  TD cohort: To define the pattern of radiological response according to MRI parameters and to correlate it with CBR and Brief Pain Inventory (BPI) parameters.
Progression-free survival - cohort 1 | 3 months
  TD cohort: To estimate the efficacy of nab-paclitaxel as measured by the progression-free survival (PFS) assessed by median time.
Variation of symptoms - cohort 1 | during first year
  TD cohort: To analyze the variation of symptoms during the first year from trial enrollment in accordance with BPI and Analgesic Quantification Algorithm (AQA).
Variation of physical function - cohort 1 | during first year
  TD cohort: To analyze the variation of physical function during the first year from trial enrollment in accordance with sponsor form.
Safety profile of nab-paclitaxel - cohort 1 | up to 12 months
  TD cohort: To evaluate the safety profile of nab-paclitaxel according to CTCAE 4.0.
Safety profile of nab-paclitaxel - cohort 2 | up to 12 months
  DSRCT and SE cohort: To evaluate the safety profile of nab-paclitaxel according to CTCAE 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martin Broto, MD, Study Director — Hospitales Universitarios Virgen del Rocío; Jaume Mora, MD, Study Director — Hospital Sant Joan de Deu; Javier Martínez Trufero, MD, Principal Investigator — Hospital Miguel Servet; Francisco Bautista, MD, Principal Investigator — Hospital Universitario Niño Jesús; Antonio López Pousa, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Roberto Díaz, MD, Principal Investigator — Hospital Universitario La Fe; José Antonio López-Martín, MD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (7):
- Spain (7):
  - H. de la Santa Creu i Sant Pau, Barcelona
  - H. Sant Joan de Déu, Barcelona
  - H.U. 12 de Octubre, Madrid
  - H.U.Niño Jesús, Madrid
  - H.U. Virgen del Rocío, Seville
  - H.U i Politècnic La Fe, Valencia
  - H.U. Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided